CLINICAL TRIAL: NCT06647134
Title: A Qualitative Assessment of the Severity and Impact of Rheumatic Immune-Related Adverse Events Following Immune Checkpoint Inhibitor Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0342; NCI-2024-07031 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Arthritis; Polymyalgia Rheumatica; Immune Checkpoint Inhibitors
Keywords: arthritis; polymyalgia rheumatica; immune related adverse events
MeSH Terms: conditions — Arthritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To understand the severity and nature of participants experiences during irAEs following immune checkpoint inhibitor immunotherapy.

DETAILED DESCRIPTION:
1. To understand the severity and nature of participants experiences during rheumatic immune-related adverse events following immune checkpoint inhibitor immunotherapy, including their functional impact
2. To explore domains relevant to participants experiencing rheumatic immune-related adverse events following immune checkpoint inhibitor immunotherapy, and attitudes to domains identified from the literature

ELIGIBILITY:
Inclusion Criteria

The criteria are:

* Patients aged 18 years and above
* English (conversational level) speaking, with the ability to give informed consent
* Patients with a rheumatologist clinician diagnosis of inflammatory arthritis irAE or PMR irAE following ICI therapy

Exclusion Criteria

* Acutely life-threatening or worsening cancer
* Hearing impairment functionally limiting participation in verbal interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Y. Jeff Li, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org